CLINICAL TRIAL: NCT00517322
Title: Left Atrial Remodelling in Hypertension: Effects of Ramipril or Irbesartan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1112
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Left Atrial Volume; Hypertensive Heart Disease; Antihypertensive Drugs; Diastolic Function; Renin Angiotensin System
Keywords: left atrial volume; hypertension; ramipril; irbesartan; diastolic function
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): treatment with ramipril
  Interventions: Drug: ramipril
- 2 (Experimental): treatment with irbesartan
  Interventions: Drug: irbesartan

INTERVENTIONS:
Drug: ramipril — ramipril 2.5- 5 mg once daily
  Arms: 1
Drug: irbesartan — irbesartan 150-300 mg once daily
  Arms: 2

SUMMARY:
Aim of the study is to compare in hypertensive patients the effect of one year therapy with ACE-inhibitor (RAMIPRIL) or angiotensin II receptor blocker (IRBESARTAN) on left atrial remodelling and diastolic function.

ELIGIBILITY:
Inclusion Criteria:·

* mild to moderate essential hypertension
* no antihypertensive treatment
* good quality echocardiogram

Exclusion Criteria:

* cardiovascular diseases (AMI, stroke o TIA)
* heart failure, valvular heart disease
* diabetes
* secondary hypertension
* atrial fibrillation
* hepatic and renal severe failure
* pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-08; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
left atrial volume | one year
diastolic function | one year

SECONDARY OUTCOMES:
systolic and diastolic blood pressure | one year

CONTACTS AND LOCATIONS:
Overall Officials: anna maria grandi, MD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- University of Insubria-Department of Clinical Medicine, Varese, Italy

REFERENCES:
- [Background] Matsuda M, Matsuda Y. Mechanism of left atrial enlargement related to ventricular diastolic impairment in hypertension. Clin Cardiol. 1996 Dec;19(12):954-9. doi: 10.1002/clc.4960191211. PMID 8957600
- [Background] Tsang TS, Barnes ME, Gersh BJ, Bailey KR, Seward JB. Left atrial volume as a morphophysiologic expression of left ventricular diastolic dysfunction and relation to cardiovascular risk burden. Am J Cardiol. 2002 Dec 15;90(12):1284-9. doi: 10.1016/s0002-9149(02)02864-3. PMID 12480035
- [Background] Healey JS, Baranchuk A, Crystal E, Morillo CA, Garfinkle M, Yusuf S, Connolly SJ. Prevention of atrial fibrillation with angiotensin-converting enzyme inhibitors and angiotensin receptor blockers: a meta-analysis. J Am Coll Cardiol. 2005 Jun 7;45(11):1832-9. doi: 10.1016/j.jacc.2004.11.070. PMID 15936615
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782